CLINICAL TRIAL: NCT03238976
Title: Nature Sounds as a Pain and Anxiety Reducing Strategy in Patients Undergoing Breast Core Biopsy: A Randomized Study
Brief Title: Nature Sounds as a Pain and Anxiety Reducing Strategy in Patients Undergoing Breast Core Biopsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB17-0355
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: breast core biopsy; core needle biopsies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature sounds exposure (Experimental): Patients will be randomly assigned to either the nature sounds group or the standard care group.
  Patients in the nature sounds group will be exposed to continuous nature sounds during the core needle biopsy (CNB) procedure.
  The CNB procedure will continue as planned with nature sounds playing instead of the supportive dialogue. All sounds will be played out of a speaker situated in the corner of the room.
  Interventions: Other: Nature sounds
- Standard care (supportive dialogue) (No Intervention): Patients will be randomly assigned to either the nature sounds group or the standard care group.
  The CNB procedure will continue as planned with supportive dialogue which will be played out of a speaker situated in the corner of the room. This group follows the current standard of care.

INTERVENTIONS:
Other: Nature sounds — Nature sounds will be played for patients in the nature sounds exposure group.
  Arms: Nature sounds exposure

SUMMARY:
Patients will be randomly assigned to one of two groups: the group exposed to NS, or the standard care group exposed to supportive dialogue. Patients assigned to the former group will be exposed to continuous NS throughout the CNB procedure.

DETAILED DESCRIPTION:
For stereotactic biopsies, the experiment consists of six different parts: (1) A baseline 5 min biopsy planning period during which only imaging occurs after patient positioning and breast compression is complete, (2) One 2-min local anesthesia administration period during which the skin is injected with local anesthetic and an incision is made to insert the biopsy needle into the breast occurs ("stressor 1"), (3) One 2-minute post local anesthesia administration period during which imaging is obtained to confirm the position of the needle with respect to the target, (4) One 1-minute sampling period when the breast tissue is sampled ('stressor 2"), (5) One 2-minute post-CNB period, during which adequacy of obtained samples is confirmed and the need for additional sampling determined, and (6) One 2-minute period during which a biopsy marker clip is deployed and pressure dressing placed on the biopsy site.

For ultrasound biopsies, the experiment also consists of six different parts: (1) A baseline 5 min biopsy planning period during which only imaging occurs after patient is positioning, (2) One 2-min local anesthesia administration period during which local anesthesia is given at the site of biopsy and a skin incision performed ("stressor 1"), (3) One post local anesthesia administration period during which intra-procedure imaging and confirmation of adequate targeting occurs, (4) One 1-minute first-pass sampling period ('stressor 2") during which the biopsy device is advanced to the target for the first time and fired to acquire the first tissue sample, and (5) One 2-minute post-CNB period, following the first needle pass while sample adequacy is visually assessed and additional intra-procedure imaging occurs, (6) One 2-minute post-CNB period, during which a biopsy marker clip is deployed and pressure dressing placed on the biopsy site.

The total time for a single site CNB is approximately 30 minutes when performed under US-guidance, and 30-45 minutes when performed under stereotactic guidance. The added physiological recordings for this experiment are not expected to significantly prolong the duration of CNB procedures.

ELIGIBILITY:
Inclusion Criteria:

* 1) ≥ 21 years old
* 2) present for CNB
* 3) to be able to read and speak English
* 4) provide written informed consent.

Exclusion Criteria:

-

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measure of psychologic stress of patients and staff | From the start of procedure until the end, not to exceed 2 years.
  Patients and staff will be required to complete a questionnaire. Questions are organized so to capture levels of psychologic stress. The answers will be compared across the two groups and descriptive statistics will be calculated.
Measure of physiologic stress of patients and staff | From the start of procedure until the end, not to exceed 2 years.
  Parasympathetic activity will be measured by HF HRV in patients and staff. Descriptive statistics from these measurements will be calculated and compared across the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kirti Kulkarni, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States